CLINICAL TRIAL: NCT00909506
Title: Efficacy and Safety of Adjuvant Metformin for Operable Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: adjuvant metformin for BC
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2010-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Metformin 500 mg/d (Active Comparator): Metformin 500 mg/d
  Interventions: Drug: Metformin
- Metformin 1000 mg/d (Active Comparator): Metformin 1000 mg/d
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebo — Control: Receive placebo pill once every evening on 1~2 weeks.
  Receive placebo pill in every morning and evening on 3~24 weeks (twice a day).
  Arms: Placebo
Drug: Metformin — Metformin 500 mg/d: Receive oral metformin 500 mg dose once daily on 1~2 weeks.
  Receive placebo pill in every morning and oral metformin 500 mg in every evening on 3~24 weeks.
  Arms: Metformin 500 mg/d
Drug: Metformin — Metformin 1000 mg/d : Receive oral metformin 500 mg dose once daily on 1~2 weeks. (Dose-escalate)
  Receive oral metformin 500 mg in every morning and evening on 3~24 weeks (metformin 500 mg * twice a day = 1000 mg per day).
  Arms: Metformin 1000 mg/d

SUMMARY:
The investigators hypothesize that adjuvant metformin use in breast cancer patients with overweight or pre-diabetes mellitus (DM) may improve their body condition including weight loss.

In this study, the investigators aim to test the efficacy and safety of adjuvant metformin for operable breast cancer patients with overweight or pre-DM.

ELIGIBILITY:
Inclusion Criteria:

* Operable Breast cancer patients with BMI ≥ 23 or 100 ≤ FBS < 126
* From 6 month to 2 years since breast cancer operation and at least 4 weeks since chemotherapy or radiotherapy
* No drug use except Tamoxifen
* Normal OTPT & Serum creatinine (<=ULN)
* ECOG performance status 0-2 or Karnofsky PS 60-100%
* Life expectancy > 12
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Pregnancy(-) & without plan for pregnancy
* Sign a written informed consent form

Exclusion Criteria:

* Type I or II DM or concurrent use of DM control agents
* Prior use of Metformin
* Hypoglycemia (FBS< 70 with clinical symptom)
* Concurrent investigational or commercial agents
* Other diet or drug intervention for weight loss
* Concurrent use of steroid
* Abnormal liver and/or renal function
* Symptomatic congestive heart failure / Cardiac arrhythmia / Angina pectoris
* Ongoing or active infection
* lactic acidosis
* Pregnancy or ongoing breast feeding
* Anorexia, bulimia, nausea due to other disease for longer than 1 month
* Allergies or allergic reactions attributed to oral medications
* Inability to swallow or digest oral medications
* Physical or psychiatric illness that would limit compliance with study protocol
* Participants in other clinical trial

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wonshik Han, M.D., Ph.D., Principal Investigator — Department of General Surgery, Seoul National University College of Medicine & Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea